CLINICAL TRIAL: NCT07119242
Title: Evaluate the Diagnostic Efficacy, Pharmacokinetics and Safety of 68Ga-DOTATATE Injection PET/CT in NETs
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: HTA Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: YZGK-ZLYT-2023-Ⅲ-Ga
Record Dates: First submitted 2024-09-13; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: NETs
MeSH Terms: interventions — gallium Ga 68 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-DOTATATE Injection (Experimental)
  Interventions: Drug: 68Ga-DOTATATE Injection

INTERVENTIONS:
Drug: 68Ga-DOTATATE Injection — The eligible subjects who participate in 68Ga study will be intravenously injected with 68Ga-DOTATATE Injection on Day1，and undergo PET/CT examination within 60 minutes after injection. Corresponding safety examination is performed before administration of 68Ga-DOTATATE Injection, 3h±1.0h after administration, and Day2. Telephone safety visit is conducted at Day7 after administration.

SUMMARY:
Evaluate the diagnostic efficacy, pharmacokinetics and safety of 68Ga-DOTATATE injection PET/CT in NETs

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old, no gender limit;
2. Karnofsky status score >50 points;
3. Expected survival time >3 months;
4. Those who have a history of neuroendocrine tumors,but require PET/CT examination for structure, location and function evaluation and disease management, and have measurable lesions; CT, MRI, 18F-FDG PET/CT or other imaging examinations are suspected of being NETs or those with space-occupying lesions and at least one of the following:

   ① Biochemical and tumor biomarkers results of blood or urine suggest that the subject is suspected of suffering from NETs (chromogranin A,neurospecific enolase,vasoactive intestinal peptide, serotonin (urinary 5-HIAA), gastrin, somatostatin,catecholamines,calcitonin,fasting insulin,C-Peptides(proinsulin) orglucagon abnormal biochemical indicators related to neuroen docrine tumors);

   ②Multiple endocrine neoplasia type 1 (MEN1) and Lindau syndrome (VHL) with familial tendency to be susceptible to NETs (symptomatic and/or asymptomatic cases; with biochemical or anatomical imaging evidence of the disease);
5. The subjects or their guardians fully understand the content,process and possible risks of the trial and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Known to be allergic to any components or excipients of 68Ga-DOTATATE injection;
2. Unable to remain relatively still during the imaging examination (such as coughing, severe arthritis, etc.), or body shape and/or weight exceeds the applicable range of the examination equipment;
3. Unable to complete the imaging examination specified in the plan due to claustrophobia,radiation phobia or personal wishes;
4. With a history of concurrent active infection or severe heart disease;
5. Those who have used long-acting somatostatin analogs within 28 days or short-acting somatostatin analogs within 2 days before the scheduled PET/CT examination of 68Ga-DOTATATE injection;
6. Those who receive long-term and repeated treatment with high-dose glucocorticoids;
7. Pregnant or lactating women,or those who do not agree to take effective contraceptive measures from the date of signing the informed consent form to 3 months after administration;
8. Blood test results

   a) WBC: < 2 x 109/L, b) Haemoglobin:< 8.0 g/dL, c) Platelets: s 50 x 109/L, d) ALT. AST. AP:> 5 times ULN, e) Bilirubin:> 3 times ULN, f) Serum creatinine:> 1.5 times ULN
9. Those who have participated in other interventional clinical trials or are participating in other interventional clinical trials within 1 month or 5 drug half-lives( whichever is longer ) before the date of signing the informed consent,or have participated in clinical trials of radioactive drugs within 1 year before the date of signing the informed consent, and the withdrawal time is less than 3 months until the date of signing the informed consent;
10. Investigators considered unsuitable to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity at the subject level | Within 28 days following 68Ga-DOTATATE injection PET/CT in NETs
  The sensitivity and specificity at the subject level Sensitivity = Number of true positive/(Number of true positive + Number of false negative) Specificity = Number of true negative/(Number of true negative + Number of false positive)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China